CLINICAL TRIAL: NCT04718298
Title: Laparoscopic Fixation Free Obliteration of Inguinal Hernia Defect With the 3D Dynamic Responsive Implant ProFlor-E - Feasibility Study
Brief Title: Laparoscopic Hernia Defect Obliteration With ProFlor-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giuseppe Amato, Consultant Professor, University of Cagliari
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopic ProFlor approach
Record Dates: First submitted 2020-07-15; First posted 2021-01-22 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Laparoscopic inguinal hernia repair; Inguinal hernia defect obliteration; Fixation free hernia repair; Regenerative scaffolds
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Inguinal hernia repair laparoscopic (Experimental): recurrent inguinal hernia after open repair or bilateral hernia patients
  Interventions: Device: ProFlor laparoscopic technique

INTERVENTIONS:
Device: ProFlor laparoscopic technique — Inguinal hernia repair laparoscopic

SUMMARY:
This feasibility study highlights the features of the 3D dynamic responsive prosthesis ProFlor-E® for fixation free obliteration of inguinal hernia defect

DETAILED DESCRIPTION:
The 3D dynamic-responsive prosthesis for inguinal hernia repair ProFlor-E® recently introduced to the market has been laparoscopically employed for the repair of one recurrent inguinal hernia previously managed with anterior open approach. The scope of this feasibility study is to demonstrate that the positive effects of the 3D implant already proven in open inguinal hernia repair are also effective or even superior for the laparoscopic of recurrent/bilateral inguinal hernias compared to conventional treatment concept.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent inguinal hernia already repaired with open approach or suffering by bilateral inguinal hernias

Exclusion Criteria:

* ASA >4 patients

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of inguinal hernia defect obliteration with ProFlor | intraoperative
  Effectiveness of the laparoscopic procedure for inguinal hernia repair with ProFlor

SECONDARY OUTCOMES:
Postoperative pain | from early stage until 18 months postop
  assessment of postoperative pain through Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Amato, MD, Principal Investigator — University of Cagliari - University of Palermo
Locations (1):
- University of Palermo, Palermo, Please Select, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato G, Lo Monte AI, Cassata G, Damiano G, Romano G, Bussani R. A new prosthetic implant for inguinal hernia repair: its features in a porcine experimental model. Artif Organs. 2011 Aug;35(8):E181-90. doi: 10.1111/j.1525-1594.2011.01272.x. Epub 2011 Jul 13. PMID 21752035
- [Background] Amato G, Romano G, Agrusa A, Marasa S, Cocorullo G, Gulotta G, Goetze T, Puleio R. Biologic response of inguinal hernia prosthetics: a comparative study of conventional static meshes versus 3D dynamic implants. Artif Organs. 2015 Jan;39(1):E10-23. doi: 10.1111/aor.12416. PMID 25626584
- [Background] Amato G, Romano G, Goetze T, Cicero L, Gulotta E, Calò PG, Agrusa A Fixation free inguinal hernia repair with the 3D dynamic responsive prosthesis ProFlor: Features, procedural steps and long-term results. International Journal of Surgery Open 2019; 21:34-4